CLINICAL TRIAL: NCT01690676
Title: The Effect of an Apple Polyphenol Extract Rich in Epicatechin and Flavan-3-ol Oligomers (Evesse™ EPC) on Brachial Artery Flow-mediated Vasodilatory Function (FMD)in Volunteer Subjects
Brief Title: Effect of an Apple Polyphenol Extract on Brachial Artery Flow-mediated Vasodilatory Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Danisco (Industry)
Collaborators: University of Turku (Other); 4Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Epi2012
Record Dates: First submitted 2012-09-14; First posted 2012-09-24 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Borderline Hypertension
Keywords: FMD; epicatechin; apple polyphenol; borderline hypertension
MeSH Terms: interventions — Catechin; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epicatechin (Active Comparator): The subjects will receive the study product and corresponding placebo once a day for 4 weeks in randomised order. There will be a four to five-weeks wash-out between the treatment periods.
  Interventions: Dietary Supplement: Epicatechin
- Microcrystalline cellulose (Placebo Comparator): The subjects will receive the study product and corresponding placebo once a day for 4 weeks in randomised order. There will be a four to five-weeks wash-out between the treatment periods.
  Interventions: Dietary Supplement: Microcrystalline cellulose

INTERVENTIONS:
Dietary Supplement: Epicatechin
  Arms: Epicatechin
Dietary Supplement: Microcrystalline cellulose
  Arms: Microcrystalline cellulose

SUMMARY:
Effect of apple polyphenols on FMD.

DETAILED DESCRIPTION:
The aim of this single centre, repeated-dose, double-blind, placebo-controlled, crossover study is to test the hypothesis that an orally ingested apple polyphenol extract rich in epicatechin and flavan-3-ol oligomers improves brachial artery endothelium-dependent vasodilation function (FMD) in volunteer subjects with borderline hypertension. FMD and endothelium-independent nitrate-mediated vasodilatation (NMD) of the left brachial artery will be investigated with ultrasonography at the start and end of both treatment periods. Biomarkers of vascular function and epicatechin (and metabolite) concentrations will be determined from blood samples taken at the start and end of both treatment periods. Diet diary data will be collected for the evaluation of the possible effects of diet on the study results. Adverse events data will be collected throughout the study. Safety laboratory determinations will be performed at the last visit of both treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Borderline hypertension
* Otherwise healthy
* Aged 40-65 years (inclusive)
* Not consuming high amounts (over 20 mg daily) of flavonoids

Exclusion Criteria:

* BMI >32 kg/m2
* Total serum cholesterol ≥ 8 mmol/l
* Any abnormal safety laboratory parameter or abnormal finding in ECG evaluated to be clinically significant
* Coronary artery disease
* Pregnancy or lactating
* Alcohol abuse as evaluated by medical history
* Regular smoking/using nicotine products
* Diabetes mellitus
* Apple allergy
* Use of lipid lowering medications
* Regular use of any medication that is known or believed to affect endothelial function or blood vessel constriction
* Any other condition or medication that in the opinion of the investigator would interfere with the evaluation of the study results or constitute a health risk for the subject
* High consumption of vitamin products, herbal remedies or products containing flavonoids

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Brachial flow-mediated dilation test (FMD) | At first visits of both periods baseline FMD will be recorded followed by FMD recording 1.5 hours after first dose. After 4 weeks intervention, at last visits of both periods FMD will be recorded, last dose will be taken and FMD recorded 1.5 hours after.
  ultrasonography, FMDmax%

SECONDARY OUTCOMES:
Nitrate-mediated vasodilatation response (NMD) | At the first and last visits of both periods, approximately 10 minutes after FMD.
  ultrasonography, NMDmax%
Circulating biomarkers of vascular function | Once at the first visit of both periods and once at the last visit of both periods. Blood sampling prior to the morning dose and appr. 2 h thereafter
  depends on the biomarker
BP | Once at the first visit of both periods and once at the last visit of both periods. Blood pressure will be recorded twice prior to the morning dose.
Plasma epicatechin concentration | At the first visit of both periods and at the last visit of both periods. Blood sampling prior to the morning dose and appr. 2 h thereafter
  HPLC

CONTACTS AND LOCATIONS:
Overall Officials: Kirsti Tiihonen, PhD, Study Director — Danisco; Olli Raitakari, MD, Principal Investigator — University of Turku, Turku, Finland, The Research Centre of Applied and Preventive Cardiovascular Medicine; Pia Salo, MD, PhD, Principal Investigator — University of Turku, Turku, Finland, The Research Centre of Applied and Preventive Cardiovascular Medicine; Anne Lithonius, Principal Investigator — Clinical Research Services Turku; Mika Scheinin, MD, PhD, Study Chair — Clinical Research Services Turku; Jari Turunen, MSc, Principal Investigator — 4Pharma Ltd.
Locations (1):
- University of Turku, Turku, Finland

REFERENCES:
- [Derived] Saarenhovi M, Salo P, Scheinin M, Lehto J, Lovro Z, Tiihonen K, Lehtinen MJ, Junnila J, Hasselwander O, Tarpila A, Raitakari OT. The effect of an apple polyphenol extract rich in epicatechin and flavan-3-ol oligomers on brachial artery flow-mediated vasodilatory function in volunteers with elevated blood pressure. Nutr J. 2017 Oct 27;16(1):73. doi: 10.1186/s12937-017-0291-0. PMID 29078780